CLINICAL TRIAL: NCT03753100
Title: Periprosthetic Bone Remodeling in Femoral Neck Fracture Patients: a 5-year Follow up Study Addressing the Influence of Surgical Approach on Periprosthetic Bone Mineral Density.
Brief Title: Periprosthetic Bone Remodeling in Femoral Neck Fracture Patients; a 5-year Follow up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Stein Ugland
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2018-11

CONDITIONS: Bone Mineral Density; Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periprosthetic BMD; anterolateral approach (Active Comparator): Periprosthetic bone mineral density will be measured using a DXA scanner from GE Lunar Prodigy. The initial scan was performed post-operatively during hospitalization
  Interventions: Other: Dual-energy X-ray absorbtiometry to evaluate periprosthetic bone mineral density around an uncemented stem implanted using either lateral or anterolateral approach to the hip joint
- Periprosthetic BMD; lateral approach (Active Comparator): Periprosthetic bone mineral density will be measured using DXA scanner from GE Lunar Prodigy.The initial scan was performed post-operatively during hospitalization.
  Interventions: Other: Dual-energy X-ray absorbtiometry to evaluate periprosthetic bone mineral density around an uncemented stem implanted using either lateral or anterolateral approach to the hip joint

INTERVENTIONS:
Other: Dual-energy X-ray absorbtiometry to evaluate periprosthetic bone mineral density around an uncemented stem implanted using either lateral or anterolateral approach to the hip joint — The measurement will start in the area about 2 cm proximal to the greater trochanter and will stop slightly below the tip of the prosthesis. This is the baseline scan and will be carried out twice with the patient lying on the table, but with movement between each scan. This is done to calculate the CV, Coefficient of Variation. We will use the formula from Wilkinson and associates, where delta is standard deviations (SD) of the difference between the two BMD measurements for each patient. BMD has been measured at baseline, 3 and 12 months. A DXA scan is now planned at 60 months. Changes in BMD related to the 7 Gruen zones will be registered.

SUMMARY:
Periprosthetic bone remodeling in femoral neck fracture patients: a 5-year follow up study addressing the influence of surgical approach on periprosthetic bone mineral density.

DETAILED DESCRIPTION:
Between January 2014 and July 2017 a RCT was conducted at Sorlandet Hospital Kristiansand, Norway. The trial was approved by the regional ethics committee (2013/1853/REK) and registered at ClinicalTrials.gov (ClinicalTrials.gov Identifier NCT02028468).Patients between 70 and 90 years of age with displaced femoral neck fractures, intact cognitive function and the ability to walk with or without a walking aid prior to falling were asked for their agreement to be enrolled and partition occurred after informed consent.A subgroup analysis looking at periprosthetic bone mineral density around the femoral component was part of this level 1 single-center randomized trial. 51 patients were enrolled in this DEXA study, and future examination of bone remodeling in these patients is now planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 70 and 90 years of age with displaced femoral neck fractures
* Intact cognitive function
* Ability to walk with or without a walking aid prior to falling.

Exclusion Criteria:

* Dementia
* Fractures in pathologic bone
* Patients not belonging to the hospital community
* Patients with sepsis or local infection
* Fracture not eligible to be treated with a hemiarthroplasty

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Periprosthetic bone mineral density measured by dual-energy X-ray absorbtiometry | 5-year follow- up study
  Change in bone mineral density

CONTACTS AND LOCATIONS:
Overall Officials: Glen Haugeberg, MD,PhD, Principal Investigator — Department of Rheumatology, Sorlandet hospital, Kristiansand, Norway
Locations (1):
- Departement of Orthopaedics, Sorlandet Hospital, Kristiansand, Norway

REFERENCES:
- [Derived] Ugland SH, Ugland TO, Haugeberg G, Pripp AH, Nordsletten L. Periprosthetic bone mineral density, assessed using dual energy x-ray absorptiometry, following arthroplasty in patients with femoral neck fracture: 5-year outcomes of a randomized controlled trial. J Int Med Res. 2024 Sep;52(9):3000605241276491. doi: 10.1177/03000605241276491. PMID 39268760